CLINICAL TRIAL: NCT02823041
Title: Enhancing Cognitive Training Through Exercise Following a First Schizophrenia Episode
Acronym: CT&E-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH110544 (NIH)
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: cognitive training; aerobic exercise; neurotrophic factors; randomized controlled trial; functional outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Training; Cognitive Remediation; Exercise; Case Management; Palliative Care; Employment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training & Exercise (Experimental): This arm involves a combination of systematic computerized cognitive training plus 150 minutes per week of aerobic exercise. All participants will also receive individual case management and supportive psychotherapy as well as Individual Placement and Support.
  Interventions: Behavioral: Cognitive Training; Behavioral: Aerobic Exercise; Behavioral: Case management and supportive psychotherapy; Behavioral: Individual Placement and Support
- Cognitive Training (Active Comparator): This arm includes the same systematic computerized cognitive training as the experimental condition, but without the additional aerobic exercise. All participants will also receive individual case management and supportive psychotherapy as well as and Individual Placement and Support.
  Interventions: Behavioral: Cognitive Training; Behavioral: Case management and supportive psychotherapy; Behavioral: Individual Placement and Support

INTERVENTIONS:
Behavioral: Cognitive Training — 24 weeks of systematic computerized cognitive training, 4 hours per week. The first 12 weeks involves neurocognitive training, using auditory training exercises from Posit Science Brain HQ. The 2nd 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. A weekly one-hour Bridging Skills Group is designed to aid generalization of training to everyday life situations.
  Other Names: cognitive remediation
Behavioral: Aerobic Exercise — Aerobic exercise occurs as two 45-minute sessions at the clinic and two 30-minute sessions at home weekly. Exercise involves an adaptation of interval training, including a variety of calisthenics that can be done without specialized equipment. Intensity of aerobic exercise is tailored to maintain an individualized target heart rate zone and is monitored by a heart rate recorder.
  Other Names: physical exercise
  Arms: Cognitive Training & Exercise
Behavioral: Case management and supportive psychotherapy — An individual therapist will provide weekly case management and therapy targeting the individual psychological problems and everyday functioning needs of the patient
Behavioral: Individual Placement and Support — An job/school specialist will use the Individual Placement and Support model to help participants return to school or work and provide ongoing outreach support.
  Other Names: supported education/employment

SUMMARY:
This is a confirmatory randomized controlled trial of the efficacy of a novel intervention combining neuroplasticity-based cognitive training with aerobic exercise, compared to the same systematic cognitive training alone. Treatment occurs for 6 months after randomization, with a followup assessment at 12 months. The investigators hypothesize that combining neuroplasticity-based computerized cognitive training and neurotrophin-enhancing physical exercise will produce neurotrophin increases and cognitive and functional improvements, even relative to cognitive training alone. The investigators target the period shortly after a first episode of schizophrenia to maximize the generalization of cognitive improvement to functional outcome, before chronic disability is established.

DETAILED DESCRIPTION:
The Cognitive Training and Exercise intervention consists of 24 weeks of systematic computerized cognitive training, 4 hours per week, plus aerobic exercise, 150 minutes per week. The Cognitive Training Intervention includes the same systematic cognitive training. The first 12 weeks involve neurocognitive training, using training exercises from Posit Science Brain HQ. The second 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. Aerobic exercise occurs as two 45-minute sessions at the clinic and two 30-minute sessions at home weekly. Intensity of aerobic exercise is tailored to maintain an individualized target heart rate zone and is monitored by a heart rate recorder. A weekly one-hour Bridging Skills Group with other members of the treatment condition is designed to aid generalization of training to everyday life situations. The immediate target is brain-derived neurotrophic factor. The primary treatment outcomes are overall cognitive deficit level and global functioning level.

ELIGIBILITY:
Inclusion Criteria:

1. a first episode of a psychotic illness that began within the past two years;
2. a diagnosis by DSM-5 of schizophrenia, schizoaffective disorder, mainly depressed type, or schizophreniform disorder;
3. sufficient acculturation and fluency in the English language to avoid invalidating research measures; and
4. residence likely to be within commuting distance of the UCLA Aftercare Research Program.

Exclusion Criteria:

1. inability to participate in aerobic exercise;
2. evidence of a known neurological disorder (e.g., epilepsy) or significant head injury;
3. evidence of moderate or severe alcohol or substance use disorder within the six months prior to the first episode or evidence that substance abuse triggered the psychotic episode or makes the schizophrenia diagnosis ambiguous; or
4. mental retardation, i.e. estimated premorbid IQ less than 70.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) overall composite score | 6 months
  The Overall Composite score from the MCCB is a summary of cognitive performance across seven domains.
Global Functioning Scale: mean of Role and Social ratings | 6 months
  A 10-point rating scale to evaluate role and social functioning
Brain-derived neurotrophic factor (BDNF) | 6 months
  BDNF is a key neurochemical factor known to mediate the effects of exercise in the brain

SECONDARY OUTCOMES:
YMCA fitness test | 6 months
  Cardiorespiratory fitness and muscular endurance measured by the YMCA fitness test
VO2 Max | 6 months
  A cardiovascular fitness measure derived from a treadmill test protocol
Role Functioning Scale | 6 months
  7-point ratings of Work Productivity, Independent Living, Social Relationships, Family Relationships

CONTACTS AND LOCATIONS:
Overall Officials: Keith Nuechterlein, Ph.D., Principal Investigator — UCLA Department of Psychiatry & Biobehavioral Sciences
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After primary results have been published, de-identified data for primary outcome variables will be available for sharing.

REFERENCES:
- See also: Summary of this study and others at the UCLA Aftercare Research Program — https://www.semel.ucla.edu/aftercare